CLINICAL TRIAL: NCT06964061
Title: An Open-label Study to Evaluate the Efficacy, Safety, Tolerability, and Biodegradation Period of PA5346 Ocular Implant, 115mcg When Administered to Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Evaluate Efficacy, Safety, Tolerability and Biodegradation of PA5346 Ocular Implant in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATA-CS104
Record Dates: First submitted 2025-03-18; First posted 2025-05-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-04

CONDITIONS: Open Angle Glaucoma (OAG); Ocular Hypertension (OH)
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PA5436 Ocular Implant, 115mcg (Experimental): PA5436 Ocular Implant, 115mcg administered by the Investigator into the anterior chamber of the study eye through a clear corneal injection
  Interventions: Combination Product: PA5436 Ocular Implant, 115mcg

INTERVENTIONS:
Combination Product: PA5436 Ocular Implant, 115mcg — The PA5346 Ocular Implant is supplied preloaded into the needle of a single use Administration Device ready for use.

SUMMARY:
The goal of this clinical study is to learn how effective and safe is a single administration of PA5346 Ocular Implant for the reduction of intraocular pressure in adult patients with open-angle glaucoma or ocular hypertension. It will also assess how long it takes for PA5346 Ocular Implant to dissolve in the eye.

DETAILED DESCRIPTION:
This is an open-label study that will evaluate the efficacy, safety, tolerability and biodegradation of PA5346 Ocular Implant administered as a single dose at 115mcg in adults with open-angle glaucoma or ocular hypertension.

The study plans to recruit approximately 12 participants. Eligible participants will receive a single PA5346 Ocular Implant administered into the intracameral space of the study eye and followed for approximately 52 weeks at a minimum or until the implant is no longer visible in the study eye.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide informed consent and follow study instructions
* 18 years of age or older
* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
* Qualifying IOPs across 2 visits following washout of IOP-lowering medication, if applicable
* Qualifying best-corrected visual acuity BCVA using Early Treatment Diabetic Retinopathy Study (ETDRS) chart in study eye
* Qualifying corneal endothelial cell density (CEDC) in the study eye

Key Exclusion Criteria:

* Pseudoexfoliation or pigment dispersion, narrow irido-corneal drainage angles, or existing peripheral anterior synechiae in the inferior angle either eye.
* Advanced or severe glaucoma
* Disqualifying central corneal thickness in either eye
* Significant other ocular conditions that could prevent accurate assessment of IOP and corneal health
* Uncontrolled medical conditions
* Have previously received, any injectable glaucoma medication into the anterior chamber of the study eye
* Have received intravitreal injections in the study eye within the last 3 months of the Screening Visit and anticipated need for an intravitreal injection during the course of the study
* Unwilling or unable to discontinue, in either eye, soft contact lens wear at least 2 days and hard contact lens wear 1 week before scheduled study visits and on implant administration days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy: change in mean diurnal intraocular pressure in study eye | Weeks 2, 12, 26 and 52
Incidence of ocular symptoms and ocular treatment-emergent adverse events | Day 1 through study completion at least until Week 52
  Ocular safety and tolerability (AEs)

SECONDARY OUTCOMES:
Efficacy: intraocular pressure change from baseline in study eye at different diurnal time points. | Weeks 2-52

OTHER OUTCOMES:
Time to complete biodegradation of the implant assessed by gonioscopy | Day 1 through study completion at least until Week 52

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Cataract & Eye Surgery Centre, Doncaster, Victoria
  - Cerulea Pty Ltd, East Melbourne, Victoria
  - Melbourne Eye Specialists, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No